CLINICAL TRIAL: NCT01834638
Title: Long-Term Safety and Efficacy of ABT-126 in Subjects With Schizophrenia: A Double-Blind Extension Study for Subjects Completing Study M10-855
Brief Title: Long-term Safety and Efficacy of ABT-126 in Subjects With Schizophrenia: An Extension Study for Subjects Completing Study M10-855 (NCT01655680)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study endpoint in preceding base study M10-855 not met.
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-765; 2012-005661-13 (EudraCT Number)
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2014-10

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ABT-126

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABT-126 low dose (Experimental): ABT-126 low dose
  Interventions: Drug: ABT-126
- ABT-126 middle dose (Experimental): ABT-126 middle dose
  Interventions: Drug: ABT-126
- ABT-126 high dose (Experimental): ABT-126 high dose
  Interventions: Drug: ABT-126

INTERVENTIONS:
Drug: ABT-126 — capsule(s)

SUMMARY:
This is a study of ABT-126 in the treatment of cognitive impairment associated with schizophrenia (CIAS), a long-term extension study to study M10-855 (NCT01655680).

ELIGIBILITY:
Inclusion Criteria:

* The subject was randomized into Study M10-855 and completed through Week 26 in that study.
* The subject is receiving one or more antipsychotic medications.

Exclusion Criteria:

* Additional history collected during participation in Study M10-855 provides evidence that, in the investigator's judgement, the subject does not have schizophrenia.
* The subject experienced an adverse event or abnormal finding during physical examination, vital signs, laboratory profile, and/or electrocardiogram (ECG) measurements in Study M10-855 that indicates the subject is likely to become medically unstable during the current study.
* The subject is currently taking or is expected to be prescribed any excluded medication without the approval of AbbVie medical monitor.
* The subject is currently enrolled in, or plans to participate in, another interventional study during the course of this trial.

Ages: 20 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with adverse events | up to 52 weeks
Change in laboratory test results | from Day -1 to Week 52
Change in vital signs | from Day -1 to Week 52
Change in electrocardiogram (ECG) data | from Day -1 to Week 52

SECONDARY OUTCOMES:
Change in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) | from Day -1 to Week 52
  rater based interview
Change in University of California San Diego Performance-Based Skills Assessment-2 (UPSA-2ER) | from Day -1 to Week 52
  rater based interview to evaluate functioning
Change in the Positive and Negative Syndrome Scale (PANSS) | from Day -1 to Week 52
  rater based interview to assess functioning
Change in the 16-item version of the Negative Symptom Assessment Scale (NSA-16) | from Day -1 to Week 52
  rater based interview to assess symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: George Haig, PharmD, Study Director — AbbVie
Locations (51):
- United States (27):
  - Site Reference ID/Investigator# 95398, Chino, California
  - Site Reference ID/Investigator# 95381, Costa Mesa, California
  - Site Reference ID/Investigator# 95400, Escondido, California
  - Site Reference ID/Investigator# 95406, Garden Grove, California
  - Site Reference ID/Investigator# 95378, National City, California
  - Site Reference ID/Investigator# 95390, Norwalk, California
  - Site Reference ID/Investigator# 95386, Oakland, California
  - Site Reference ID/Investigator# 95391, Oceanside, California
  - Site Reference ID/Investigator# 95380, Orange, California
  - Site Reference ID/Investigator# 95395, Pico Rivera, California
  - Site Reference ID/Investigator# 95403, Riverside, California
  - Site Reference ID/Investigator# 128356, San Bernardino, California
  - Site Reference ID/Investigator# 95405, San Diego, California
  - Site Reference ID/Investigator# 95397, San Diego, California
  - Site Reference ID/Investigator# 95384, San Gabriel, California
  - Site Reference ID/Investigator# 95385, Santa Ana, California
  - Site Reference ID/Investigator# 95387, Torrance, California
  - Site Reference ID/Investigator# 95382, New Haven, Connecticut
  - Site Reference ID/Investigator# 95399, Atlanta, Georgia
  - Site Reference ID/Investigator# 95377, Marietta, Georgia
  - Site Reference ID/Investigator# 120595, Chicago, Illinois
  - Site Reference ID/Investigator# 129380, Hoffman Estates, Illinois
  - Site Reference ID/Investigator# 95379, Cedarhurst, New York
  - Site Reference ID/Investigator# 95392, Rochester, New York
  - Site Reference ID/Investigator# 95388, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 95402, DeSoto, Texas
  - Site Reference ID/Investigator# 95393, Houston, Texas
- Russia (19):
  - Site Reference ID/Investigator# 117189, Chita
  - Site Reference ID/Investigator# 117188, Kazan'
  - Site Reference ID/Investigator# 117175, Lipetsk
  - Site Reference ID/Investigator# 117159, Moscow
  - Site Reference ID/Investigator# 117183, Moscow
  - Site Reference ID/Investigator# 117182, Novosibirsk
  - Site Reference ID/Investigator# 117157, Saint Petersburg
  - Site Reference ID/Investigator# 117185, Saint Petersburg
  - Site Reference ID/Investigator# 117192, Saint Petersburg
  - Site Reference ID/Investigator# 117193, Saint Petersburg
  - Site Reference ID/Investigator# 117176, Saint Petersburg
  - Site Reference ID/Investigator# 117195, Saint Petersburg
  - Site Reference ID/Investigator# 117186, Saint Petersburg
  - Site Reference ID/Investigator# 117156, Saratov
  - Site Reference ID/Investigator# 117177, Saratov
  - Site Reference ID/Investigator# 117180, Stavropol
  - Site Reference ID/Investigator# 117181, Yaroslavl
  - Site Reference ID/Investigator# 117194, Yekaterinburg
  - Site Reference ID/Investigator# 117178, Yekaterinburg
- United Kingdom (5):
  - Site Reference ID/Investigator# 117422, Edinburgh
  - Site Reference ID/Investigator# 117423, London
  - Site Reference ID/Investigator# 117425, London
  - Site Reference ID/Investigator# 117424, Newcastle upon Tyne
  - Site Reference ID/Investigator# 117419, Oxford

REFERENCES:
- [Result] Haig G, Wang D, Othman AA, Zhao J. The alpha7 Nicotinic Agonist ABT-126 in the Treatment of Cognitive Impairment Associated with Schizophrenia in Nonsmokers: Results from a Randomized Controlled Phase 2b Study. Neuropsychopharmacology. 2016 Nov;41(12):2893-2902. doi: 10.1038/npp.2016.101. Epub 2016 Jun 20. PMID 27319970